CLINICAL TRIAL: NCT01035619
Title: A Single-Center, Open-Label, Single-Dose Study To Assess The Pharmacokinetics, Safety, And Tolerability Of Moxidectin In Subjects Aged 4 To 11 Years ( >=12 kg) With Or Without Onchocerca Volvulus Infection
Brief Title: Pediatric Pharmacokinetics And Safety Study Of Moxidectin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1751005; 3110A1-2201
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Onchocerciasis
Keywords: onchocerciasis; river blindness; moxidectin; pediatric
MeSH Terms: conditions — Onchocerciasis; Onchocerciasis, Ocular | interventions — moxidectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Moxidectin (Experimental)
  Interventions: Drug: moxidectin

INTERVENTIONS:
Drug: moxidectin — Single Dose Moxidectin 4 mg

SUMMARY:
The purpose of this study is to measure the amount of moxidectin in subjects' blood and to measure safety. This study will enroll 36 children aged 4 to 11 years (>=12 kg) with or without Onchocerca volvulus (O volvulus) infection. O volvulus is the nematode, or roundworm, that causes Onchocerciasis, also known as river blindness. Each subject will receive a single dose of 4 mg moxidectin (orally administered) and will be followed inpatient from screening through day 13 and as outpatients through month 6. The study will take place at a single research center.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 4 to 11 years, inclusive (weighing >= 12 kg)
* With or without O volvulus infection

Exclusion Criteria:

* Any major illness/condition that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in and completion of the study
* Contraindication or hypersensitivity to moxidectin

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The amount of moxidectin in subjects blood, as measured by collecting a number of blood samples from each subject, in which the amount of moxidectin will be measured | 3 months

SECONDARY OUTCOMES:
The safety and tolerability of a single dose of 4 mg moxidectin in subjects as measured by physical examinations, laboratory tests, vital signs and ECG findings | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1751005&StudyName=Pediatric%20Pharmacokinetics%20And%20Safety%20Study%20Of%20Moxidectin